CLINICAL TRIAL: NCT00690937
Title: A Multicenter, Single-blind, Active and Placebo-controlled, Parallel-group, Randomized Study of Two Dosing Regimens of Enteric Coated Sevelamer in Patients With Mild to Moderate Hypercholesterolemia
Brief Title: A Multicenter, Active and Placebo-controlled Study of Enteric Coated Sevelamer in Patients With Mild to Moderate Hypercholesteremia
Acronym: Sevelamer ECS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Manipal Acunova Ltd. (Network)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECS00107; ELLS
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia, bile acid sequestrant, LDL-cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 ECS (Experimental): Low dose treatment
  Interventions: Drug: Enteric coated sevelamer
- 2 ECS (Experimental): High dose treatment
  Interventions: Drug: Enteric coated sevelamer
- 3 Colesevelam (Active Comparator): Active control treatment
  Interventions: Drug: Colesevelam Cholestagel
- 4 Placebo (Placebo Comparator): Placebo matched to low dose treatment
  Interventions: Drug: Placebo
- 5 Placebo (Placebo Comparator): Placebo matched to high dose treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enteric coated sevelamer — Drug treatment
  Other Names: ECS
  Arms: 1 ECS
Drug: Enteric coated sevelamer — Drug treatment
  Arms: 2 ECS
Drug: Colesevelam Cholestagel — Drug comparator
  Arms: 3 Colesevelam
Drug: Placebo — Placebo
  Arms: 4 Placebo
Drug: Placebo — Placebo
  Arms: 5 Placebo

SUMMARY:
A total of 120 patients will be entered in this study to assess the safety and efficacy of enteric coated sevelamer (ECS) to lower LDL cholesterol. Patients will be randomized into two active treatment groups, two placebo groups and one active control group.

DETAILED DESCRIPTION:
This is a prospective, randomized, single blind, active and placebo-controlled, parallel-group, multi-center study.

Two groups of ECS consisting of 3 and 6 tablets/day (n=30), two placebo groups of 3 and 6 tablets/day (n=15 each) and one active control group of colesevelam 6 tablets/day (n=30). The study is being conducted solely in India and there will be a total of 6-8 sites.

The safety parameters are:

* Serious adverse events SAEs
* Treatment and non-treatment emergent AEs
* Physical exams and vital signs
* Clinical safety laboratories

The efficacy parameters include a fasting lipid profile:

* Low density lipoproteins (LDL)
* Total cholesterol
* High density lipoproteins (HDL)
* Triglycerides

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older
* Clinical diagnosis of mild to moderate hypercholesterolemia 1)LDL cholesterol greater than or equal to 130 mg/dL and less than or equal to 220 mg/dL 2) Triglycerides less than or equal to 300 mg/dL

Exclusion Criteria:

* Women who are pregnant or lactating.
* Patients using other lipid-lowering medications during .
* Patients with unstable medical conditions and/or comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoints are: The type and number of AEs and proportion of patients with AEs. | throughout study
Assessment of clinical laboratory parameters including blood chemistry, liver function tests, and renal function tests and hematology (CBC). | throughout study
The primary efficacy endpoint is: The percent change in LDL cholesterol from baseline. | From baseline to Day 42

SECONDARY OUTCOMES:
The secondary efficacy endpoints are: the absolute change in LDL cholesterol from baseline. | From baseline to Day 42
The percent change in total cholesterol, HDL cholesterol and triglycerides from baseline. | From baseline to Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- India (8):
  - Diacon Hospital and Research Center, Bangalore
  - M S Ramaiah Medical College and Memorial Hospital, Bangalore
  - Appollo first Med Hospital, Chennai
  - Associates in Clinical Endocronolgy Education & Research (ACEER), Chennai
  - Care Hospital, Hyderabad
  - Diabetes Endocrine Nutrition Management and Research Center, Mumbai
  - P D Hinduja National Hospital and Medical Research Centre, Mumbai
  - Indraprastha Apollo Hospitals, New Delhi